CLINICAL TRIAL: NCT03345056
Title: Evaluation of Vitrectomy With Planned Foveal Detachment as Surgical Treatment for Refractory Diabetic Macular Edema With or Without Vitreo-macular Interface Abnormality
Brief Title: Vitrectomy With Planned Foveal Detachment for Refractory DME With or Without Vitreo-macular Interface Abnormality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, ahmed M. Abdel hadi, Assistant professor of ophthalmology, Ministry of Health and Population, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHEgypt
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Chronic Edema of the Macula
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- included cases (Other): vitrectomy done with planned foveal separation and followed for the result
  Interventions: Procedure: vitrectomy with planned foveal detachment

INTERVENTIONS:
Procedure: vitrectomy with planned foveal detachment — 23 gauge vitrectomy, posterior hyaloid detachment, internal limiting membrane peeling , sub-macular BSS injection using 38 gauge canula
  Other Names: vitrectomy with submacular BSS injection

SUMMARY:
To evaluate the therapeutic efficacy of sub retinal BSS injections in conjunction with conventional vitrectomy for refractory Diabetic macular edema (DME)- resistant to more than one anti-VEGF agent, intravitreal corticosteroids and to previous vitrectomy. Some of enrolled cases had normal vitreo-macular interface (VMI) relationship, while other cases had incomplete vitreoretinal separation with vitreomacular attachment (VMA).

ELIGIBILITY:
Inclusion Criteria:

* Cases with refractory DME with a central macular thickness (CMT) of more than 300 µm despite undergoing anti-VEGF therapy (5-6 monthly injections of ranibizumab (IVR) or bevacizumab (IVB) with shifting to aflibercept (IVA) for additional 3 injections).

Exclusion Criteria:

* The major exclusion criteria were: (1) presence of apparent retinal pigment epithelium (RPE) atrophy at or near the macula; (2) presence of proliferative diabetic fibrovascular membranes threating or at the macula; (3) presence of diabetic optic atrophy; and (4) presence of neovascular glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
central macular thickness decrease | 10 months postperative
  decrease in central macular thickness by OCT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel Hadi AM. Evaluation of Vitrectomy with Planned Foveal Detachment as Surgical Treatment for Refractory Diabetic Macular Edema with or without Vitreomacular Interface Abnormality. J Ophthalmol. 2018 May 7;2018:9246384. doi: 10.1155/2018/9246384. eCollection 2018. PMID 29854429